CLINICAL TRIAL: NCT01418690
Title: Changes in Tissue Oxygenation Following Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB11-00509
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Non-invasive near infra-red device (NIRS)

SUMMARY:
Adequate tissue oxygenation is required for effective white blood cell function and bactericidal activity. Decreased tissue oxygenation is a risk factor for perioperative wound infections. Regional anesthetic techniques result in a functional sympathetic block and may increase tissue oxygenation. The purpose of this study is to evaluate changes in tissue oxygenation using a non-invasive Near-infrared spectroscopy (NIRS) device. The current study will evaluate changes in tissue oxygenation following regional anesthetic techniques (peripheral nerve blockade and neuraxial techniques such as caudal block) in pediatric patients).

Regional anesthesia will induce a sympathetic blockade and improve tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical procedure who have consented to a regional block.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring regional anesthetics.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation | 1 Day (Day of Surgery)
  NIRS values from two sites before and after the regional anesthetic is placed.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States